CLINICAL TRIAL: NCT02953210
Title: Comparative Randomized Controlled Trial Study of General Balanced Anesthesia Based on Opioid and Opioid Sparing Balanced Anesthesia for Cholecystectomy Surgery Via Laparoscopy: Intraoperative and Postoperative Outcomes
Brief Title: Laparoscopic Cholecystectomy: General Anesthesia With Opioid Versus General Opioid Free Anesthesia
Acronym: GALOFF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of São Paulo (Other)
Collaborators: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Marcelo Vaz Perez, principal investigator, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: opioid free anesthesia
Record Dates: First submitted 2016-10-26; First posted 2016-11-02 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Pain, Postoperative; Anesthesia Complication; Nausea; Vomiting; Ileus Paralytic; Hemodynamic Instability
MeSH Terms: conditions — Pain, Postoperative; Nausea; Vomiting; Ileus | interventions — Ketamine; Lidocaine; Fentanyl; Clonidine; Midazolam; Isoflurane; Rocuronium; Propofol; dexamethasone-21-sulfobenzoate; Ranitidine; Ondansetron; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GF general free (Experimental): pre induction midazolam 50ug.kg-1, clonidine 1ug.kg induction dexter ketamine 0.2mg.kg, lidocaine 1.5mg.kg, propofol 2mg.kg,rocuronium 0.6mg.kg maintenance isoflurane 1 CAM, lidocaine 2mg.kg.h
  Interventions: Drug: dexter ketamine; Drug: Lidocaine Hydrochloride; Drug: Clonidine Hydrochloride; Drug: Midazolam Hydrochloride; Drug: Isoflurane Volatile Liquid; Drug: Rocuronium Injectable Solution; Drug: Propofol 1 % Injectable Suspension; Drug: Dexamethasone-21-Sulfobenzoate, Sodium Salt; Drug: Ranitidine Hydrochloride; Drug: Ondansetron Hydrochloride; Drug: Ketorolac Injectable Solution; Drug: Bupivacaine Hydrochloride
- GBal general balanced (Active Comparator): pre induction with midazolam 50 ug.kg induction fentanyl 3ug.kg, propofol 2mg.kg, rocuronium 0.6mg.k maintenance isoflurane 1 CAM and fentanyl as needed
  Interventions: Drug: Fentanyl Hydrochloride; Drug: Midazolam Hydrochloride; Drug: Isoflurane Volatile Liquid; Drug: Rocuronium Injectable Solution; Drug: Propofol 1 % Injectable Suspension; Drug: Dexamethasone-21-Sulfobenzoate, Sodium Salt; Drug: Ranitidine Hydrochloride; Drug: Ondansetron Hydrochloride; Drug: Ketorolac Injectable Solution; Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: dexter ketamine — multimodal anesthesia without opioids ketamine as induction drug
  Other Names: ketamine plus
  Arms: GF general free
Drug: Lidocaine Hydrochloride — continuous infusion intravenous
  Other Names: xylocaine
  Arms: GF general free
Drug: Fentanyl Hydrochloride — intravenous
  Other Names: Fentanil
  Arms: GBal general balanced
Drug: Clonidine Hydrochloride — clonidine intravenous pre induction
  Other Names: Catapres
  Arms: GF general free
Drug: Midazolam Hydrochloride — premedication
Drug: Isoflurane Volatile Liquid — maintenance of general anesthesia
  Other Names: isoflurane
Drug: Rocuronium Injectable Solution — induction of general anesthesia
  Other Names: rocuronium
Drug: Propofol 1 % Injectable Suspension — induction of general anesthesia
  Other Names: propofol
Drug: Dexamethasone-21-Sulfobenzoate, Sodium Salt — at the end of the procedure 4mg IV
Drug: Ranitidine Hydrochloride — at the end of the procedure
Drug: Ondansetron Hydrochloride — at the end of the procedure
  Other Names: ondasetron
Drug: Ketorolac Injectable Solution — at the of the procedure
  Other Names: keterolac
Drug: Bupivacaine Hydrochloride — at the end of the procedure for infiltration of trocar wounds
  Other Names: bupivacaine

SUMMARY:
The use of opioid during surgery can cause side effects and may delay hospital discharge. Some studies have shown balanced sparing opioid anesthesia can optimize the side effects and and the time of discharge. In this compared controlled randomized study the aim is to evaluate the intraoperative and postoperative pain, hemodynamic effects, nausea/vomiting, postoperative ileus, sedation, urinary retention, time of discharge PACU Post anesthesia care unit and hospital.

DETAILED DESCRIPTION:
Patients under laparoscopic cholecystectomy has moderate to severe pain. This study will compare intraoperative hemodynamic parameters under two techniques of general anesthesia: The primary outcome pain was used for planning the sample size of participants and considered a variation of 3 points on VAS (Visual analogic scale of pain). The secondaries outcomes nausea/vomiting, sedation, ileus paralytics, urinary retention, time of discharge (PACU) and hospital stay, and patient satisfaction will be recorded and analyzed.

the patients will be allocated from randomized program in one of the two arms.

1. Based opioid balanced anesthesia propofol, fentanyl, rocuronium and isoflurane
2. Opioid sparing balance anesthesia with propofol, dexter- ketamine, clonidine, midazolan,isoflurane and lidocaine.

At the end of procedure both groups will receive dexamethasone, ranitidine

, ondansetron, keterolac IV and local infiltration of bupivacaine on trocar wounds as multimodal analgesia.

General anesthesia opioid free seems to have less side effects than the general anesthesia based on opioid this study will compare it.

ELIGIBILITY:
Inclusion Criteria:

* Patient under Laparoscopic cholecystectomy routine American Society of Anesthesiology ASA I or II

Exclusion Criteria:

* chronic use of opioids
* Body mass index (BMI) > 35 Kg.m-2
* Chronic heart failure, renal and hepatic failure
* illicit drugs users
* cognitive impairments

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 60min after the surgery
  will be asked pain at rest and movement and cough using the analog verbal scale of pain

SECONDARY OUTCOMES:
nausea/ vomiting | 12, 24 and 36 hours after surgery
  will be asked yes or not and how many times
Paralytic ileus | 12, 24 and 36 hours after surgery
  will be access with ultrasound movement of intestine
first analgesic rescue requirement | 12 hours after the surgery
  the first analgesic given at PACU when the patient asked for it
pruritus | 12, 24 , 36 hours after surgery
  yes or no, mild, moderate to serve
sedation | 12, 24 and 26 hours after surgery
  will be use the Ramasay scale
time of discharge of PACU | 12 hour after the surgery
  time when the patient will transfer to ward after the surgery
Hemodynamics effects | intraoperative
  mean arterial pressure
weight | Baseline
  measure in kilogram
height | Baseline
  measure in cm
gender | Baseline
  male or female
saturation of o2 | intraoperative
  oximetry
ETCO2 | intraoperative
  capnography
heart rate | intraoperative
  heart rate
pain | 12, 24 and 36 hours after the procedure
  will be asked pain at rest and movement and cough using the analog verbal scale of pain

CONTACTS AND LOCATIONS:
Overall Officials: marcelo v perez, PhD, Principal Investigator — Faculdade De Ciencias Medicas da Santa Casa de Sao Paulo
Locations (1):
- Faculdade de Ciências Médicas da Santa Casa de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bisgaard T. Analgesic treatment after laparoscopic cholecystectomy: a critical assessment of the evidence. Anesthesiology. 2006 Apr;104(4):835-46. doi: 10.1097/00000542-200604000-00030. PMID 16571981
- [Background] De Oliveira GS Jr, Fitzgerald P, Streicher LF, Marcus RJ, McCarthy RJ. Systemic lidocaine to improve postoperative quality of recovery after ambulatory laparoscopic surgery. Anesth Analg. 2012 Aug;115(2):262-7. doi: 10.1213/ANE.0b013e318257a380. Epub 2012 May 14. PMID 22584558
- [Result] Collard V, Mistraletti G, Taqi A, Asenjo JF, Feldman LS, Fried GM, Carli F. Intraoperative esmolol infusion in the absence of opioids spares postoperative fentanyl in patients undergoing ambulatory laparoscopic cholecystectomy. Anesth Analg. 2007 Nov;105(5):1255-62, table of contents. doi: 10.1213/01.ane.0000282822.07437.02. PMID 17959952